CLINICAL TRIAL: NCT02553460
Title: Total Therapy for Infants With Acute Lymphoblastic Leukemia (ALL) I
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Gateway for Cancer Research (Other); Baylor College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TINI; NCI-2015-01493 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2015-09-16; First posted 2015-09-17 (Estimated); Results first posted 2023-06-07 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Infants
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Methotrexate; Dexamethasone; Calcium Dobesilate; Mitoxantrone; pegaspargase; asparaginase erwinia chrysanthemi recombinant; Asparaginase; Bortezomib; Vorinostat; Cyclophosphamide; Mercaptopurine; Leucovorin; Cytarabine; Etoposide; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants who meet eligibility requirements will receive remission induction, consolidation treatment, reinduction, reintensification and maintenance therapy.
  Interventions: ITMHA, dexamethasone, mitoxantrone, pegaspargase or asparaginase Erwinia chrysanthemi, bortezomib, vorinostat, cyclophosphamide, mercaptopurine, methotrexate, leucovorin calcium, cytarabine, etoposide, and vincristine.
  Interventions: Drug: ITMHA; Drug: Dexamethasone; Drug: Mitoxantrone; Drug: Pegaspargase; Drug: Asparaginase Erwinia Chrysanthemi; Drug: Bortezomib; Drug: Vorinostat; Drug: Cyclophosphamide; Drug: Mercaptopurine; Drug: Methotrexate; Drug: Leucovorin Calcium; Drug: Cytarabine; Drug: Etoposide; Drug: Vincristine

INTERVENTIONS:
Drug: ITMHA — Given intrathecally (IT).
  Other Names: Intrathecal Triples; Methotrexate/hydrocortisone/cytarabine
Drug: Dexamethasone — Given orally (PO) or naso-gastrically (NG) or intravenously (IV).
  Other Names: Decadron®; Hexadrol®; Dexone®; Dexameth®
Drug: Mitoxantrone — Given IV.
  Other Names: Novantrone®; Mitozantrone
Drug: Pegaspargase — Given IV. If participant is allergic to pegaspargase, Asparaginase Erwinia Chrysanthemi will be used.
  Other Names: PEG-asparaginase; Oncaspar®
Drug: Asparaginase Erwinia Chrysanthemi — Asparaginase Erwinia Chrysanthemi will be used in case of allergy or intolerance of participant to PEG-asparaginase. Given IV (preferred) or intramuscularly (IM).
  Other Names: Erwinia chrysanthemi; Erwinase®; Erwinaze^T^M; Crisantaspase
Drug: Bortezomib — Given IV.
  Other Names: Velcade®; PS-341; MLN341; LDP-341
Drug: Vorinostat — Taken PO or NG.
  Other Names: Solinza®; Suberoylanidide Hydroxamic Acid; SAHA
Drug: Cyclophosphamide — Given IV.
  Other Names: Cytoxan®
Drug: Mercaptopurine — Given PO or NG.
  Other Names: 6-MP; Purinethol®
Drug: Methotrexate — Given IV, IM or PO.
  Other Names: MTX; High Dose MTX
Drug: Leucovorin Calcium — Leucovorin rescue PO or IV.
  Other Names: Wellcovorin®; Folinic acid
Drug: Cytarabine — Given IV.
  Other Names: Ara-C; Cytosar-U®
Drug: Etoposide — Given IV. In case of participant allergy, etoposide phosphate (Etopophos®) will be given.
  Other Names: VP-16; Vepesid®
Drug: Vincristine — Given IV.
  Other Names: Oncovin®

SUMMARY:
The purpose of this study is to test the good and bad effects of the study drugs bortezomib and vorinostat when they are given in combination with chemotherapy commonly used to treat acute lymphoblastic leukemia (ALL) in infants. For example, adding these drugs could decrease the number of leukemia cells, but it could also cause additional side effects. Bortezomib and vorinostat have been approved by the US Food and Drug Administration (FDA) to treat other cancers in adults, but they have not been approved for treating children with leukemia. With this research, we plan to meet the following goals:

PRIMARY OBJECTIVE:

* Determine the tolerability of incorporating bortezomib and vorinostat into an ALL chemotherapy backbone for newly diagnosed infants with ALL.

SECONDARY OBJECTIVES:

* Estimate the event-free survival and overall survival of infants with ALL who are treated with bortezomib and vorinostat in combination with an ALL chemotherapy backbone.
* Measure minimal residual disease (MRD) positivity using both flow cytometry and PCR.
* Compare end of induction, end of consolidation, and end of reinduction MRD levels to Interfant99 (ClinicalTrials.gov registration ID number NCT00015873) participant outcomes.

DETAILED DESCRIPTION:
Treatment will consist of 4 main phases: Remission Induction, Consolidation, Reinduction, and Maintenance. High risk patients will receive a reintensification phase prior to transplant in first remission.

REMISSION INDUCTION: Chemotherapy will be given in an attempt to induce the participant's leukemia into remission. Drugs given are intrathecal triple drug treatment with methotrexate, hydrocortisone and Ara-C (ITMHA); dexamethasone; vorinostat; bortezomib; PEG-asparaginase; mitoxantrone; cyclophosphamide; cytarabine; and 6-mercaptopurine.

CONSOLIDATION PHASE: After the participant's blood counts have recovered from Remission Induction, he/she will move to the consolidation phase. This therapy is given to kill any remaining leukemia cells. Drugs given are ITMHA, high-dose methotrexate, and 6-mercaptopurine.

RE-INDUCTION: This phase aims to improve the participant's overall response to therapy by again seeking to bring his/her leukemia into remission. Drugs given are ITMHA, mitoxantrone, peg-asparaginase, dexamethasone, bortezomib, and vorinostat.Participants that achieve MRD negative status following Re-Induction may proceed directly to stem cell transplant (SCT) (SCT not part of this study).

RE-INTENSIFICATION: Participants that remain MRD positive following Consolidation or Reinduction may receive Chimeric Antigen Receptor T-Cell therapy (CART), if available (CART is not part of this study), or proceed to a Reintensification phase then go on to stem cell transplant (SCT).

MAINTENANCE PHASE: Participants with negative MRD after consolidation will skip the re-intensification phase and proceed to receive maintenance therapy to keep the leukemia from returning. Drugs given are ITMHA, dexamethasone, vincristine, 6-mercaptopurine and methotrexate. Each cycle of these drugs lasts 28 days and will be repeated up to 20 times as long as there are no serious side effects.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≤ 365 days of age at the time of diagnosis.
* Patient has newly diagnosed acute lymphoblastic leukemia (ALL) or acute undifferentiated leukemia with ≥25% blasts in the bone marrow (M3), with or without extramedullary disease. Patients with T-cell ALL are eligible. Patients with bilineage or biphenotypic acute leukemia are eligible, provided the morphology and immunophenotype are predominantly lymphoid.
* Limited prior therapy, including hydroxyurea for 72 hours or less, systemic glucocorticoids for one week or less, one dose of vincristine, and one dose of intrathecal chemotherapy.
* Written informed consent following Institutional Review Board, NCI, FDA, and Office for Human Research Protections (OHRP) Guidelines.

Exclusion Criteria:

* Patients with prior therapy, other than therapy specified in the Inclusion Criteria.
* Patients with mature B-cell ALL or acute myelogenous (AML).
* Patients with Down syndrome.
* Inability or unwillingness of legal guardian/representative to give written informed consent.

Max Age: 365 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-01-29 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2031-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Gruber, MD, PhD, Study Chair — Lucile Packard Children's Hospital Stanford University; Sima Jeha, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (15):
- United States (9):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - Children's Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - St. Jude Affiliate-Charlotte, Charlotte, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Children's Hospital of the King's Daughters (CHKD), Norfolk, Virginia
- Canada (6):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - Children's & Women's Health Centre of British Columbia, Vancouver, British Columbia
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
  - The Montreal Children's Hospital (MUHC-McGill), Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fifty patients were enrolled between January 2016 to November 2021.
Groups:
- Stratum 1: Patient is < 365 days of age at the time of diagnosis. Patient has newly diagnosed acute lymphoblastic leukemia (ALL) or acute undifferentiated leukemia with ≥25% blasts in the bone marrow (M3), with or without extramedullary disease. Patients with T-cell ALL are eligible. Patients with bilineage or biphenotypic acute leukemia are eligible, provided the morphology and immunophenotype are predominantly lymphoid. Limited prior therapy, including hydroxyurea for 72 hours or less, systemic glucocorticoids for one week or less, one dose of vincristine, and one dose of intrathecal chemotherapy. Written informed consent following Institutional Review Board, NCI, FDA, and OHRP Guidelines.
Period: Overall Study
Arm/Group | Stratum 1
Started | 50
Completed | 27
Not Completed | 23
Not completed — Death | 3
Not completed — Withdrawal by Subject | 1
Not completed — Development of unacceptable toxicity during treatment | 1
Not completed — Relapse or Transplant | 14
Not completed — No response to treatment | 2
Not completed — CAR T cells | 2

BASELINE CHARACTERISTICS:
Arm/Group | Stratum 1
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: months] | 5.32 (3.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 31
  Black | 4
  Other | 15
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 13
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Treatment-related Mortality (TRM)
Description: Number of treatment related deaths divided by total number of patients during induction or reinduction therapy.
  Presented as percentage
Time Frame: At the end of reinduction (up to 5 months after start of therapy)
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum 1
Number analyzed (Participants) | 50
Participants | 1

2. Secondary Outcome: Percentage of Participants With 3-year Event Free Survival (EFS)
Description: Event-free survival (EFS) will be estimated by the Kaplan-Meier estimator. For EFS, relapse and second malignancies will be considered as failures in addition to death in complete remission. The time to EFS will be set to 0 for patients who fail to achieve complete remission. EFS probability will be estimated with 95% confidence intervals.
Time Frame: 3 years after completion of therapy (up to 5 years after start of therapy)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stratum 1
Number analyzed (Participants) | 50
percentage of participants | 49.96 [34.9 to 63.3]

3. Secondary Outcome: Percentage of Participants With 5-year Overall Survival (OS)
Description: Overall survival (OS) will be estimated by the Kaplan-Meier estimator with 95% confidence intervals.
Time Frame: 5 years after completion of therapy (up to 7 years after start of therapy)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stratum 1
Number analyzed (Participants) | 50
percentage of participants | 62.8 [46.6 to 75.3]

4. Secondary Outcome: Minimal Residual Disease (MRD) Positivity Using Flow Cytometry or PCR at Induction Day 22, End of Induction, End of Consolidation, and End of Maintenance.
Description: Proportion of participants with positive MRD at the end of each therapy block. The proportion of MRD positive patients is determined by the number of patients that are MRD positive at the end of each therapy block divided by the number of patients that completed each therapy block.
Time Frame: At the end of induction day 22 (approximately 3 weeks), end of induction (approximately 6 weeks), end of consolidation (approximately 14 weeks), and end of maintenance therapy (approximately 2 years)
Population: The number analyzed is different from the overall number analyzed because the patient(s) MRD at that time period was not evaluated due to induction failure, death, or relapse.
Measure: Count of Participants; unit: Participants
Arm/Group | Stratum 1
Number analyzed (Participants) | 49
Participants
  MRD positivity at Day 22 | 13
  MRD positivity at End of Induction | 13
  MRD positivity at End of Consolidation: number analyzed (Participants) | 46
  MRD positivity at End of Consolidation | 11
  MRD positivity at End of Maintenance: number analyzed (Participants) | 27
  MRD positivity at End of Maintenance | 0

ADVERSE EVENTS:
Time Frame: Adverse event data are collected from Induction day 1 until 30 days after the end of maintenance, approximately 2 years. Some patients are still receiving treatment.
Arm/Group | Stratum 1
All-Cause Mortality (participants affected / at risk) | 17/50
Serious Adverse Events (participants affected / at risk) | 27/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1 (N=50)
Febrile neutropenia (Blood and lymphatic system disorders) | 8 (14)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Heart failure (Cardiac disorders) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Myocarditis (Cardiac disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Ileal perforation (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 6 (11)
Infections and infestations - Other, specify (Infections and infestations) | 10 (15)
Lung infection (Infections and infestations) | 4 (11)
Meningitis (Infections and infestations) | 1 (1)
Peritoneal infection (Infections and infestations) | 1 (1)
Rhinitis infective (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 4 (5)
Skin infection (Infections and infestations) | 1 (1)
Small intestine infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 4 (6)
Wound infection (Infections and infestations) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (2)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 2 (2)
Seizure (Nervous system disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1 (N=50)
Anemia (Blood and lymphatic system disorders) | 49 (574)
Febrile neutropenia (Blood and lymphatic system disorders) | 29 (52)
Leukocytosis (Blood and lymphatic system disorders) | 4 (4)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 2 (2)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 2 (3)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (4)
Ascites (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 3 (3)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 13 (18)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (3)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 6 (7)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1)
Typhlitis (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 7 (15)
General disorders and administration site conditions - Other, specify (General disorders) | 3 (3)
Irritability (General disorders) | 2 (2)
Localized edema (General disorders) | 2 (2)
Pain (General disorders) | 5 (5)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 2 (2)
Abdominal infection (Infections and infestations) | 2 (2)
Catheter related infection (Infections and infestations) | 5 (7)
Enterocolitis infectious (Infections and infestations) | 14 (19)
Infections and infestations - Other, specify (Infections and infestations) | 15 (18)
Lung infection (Infections and infestations) | 7 (15)
Mucosal infection (Infections and infestations) | 5 (10)
Otitis media (Infections and infestations) | 7 (9)
Penile infection (Infections and infestations) | 1 (2)
Rhinitis infective (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 5 (8)
Upper respiratory infection (Infections and infestations) | 19 (25)
Urinary tract infection (Infections and infestations) | 7 (9)
Wound infection (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 2 (3)
Alanine aminotransferase increased (Investigations) | 40 (150)
Alkaline phosphatase increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 18 (26)
Blood bilirubin increased (Investigations) | 9 (46)
Cholesterol high (Investigations) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
Fibrinogen decreased (Investigations) | 2 (2)
GGT increased (Investigations) | 6 (12)
Investigations - Other, specify (Investigations) | 1 (14)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 48 (878)
Lymphocyte count increased (Investigations) | 9 (14)
Neutrophil count decreased (Investigations) | 50 (927)
Platelet count decreased (Investigations) | 50 (832)
Weight gain (Investigations) | 2 (9)
Weight loss (Investigations) | 7 (11)
White blood cell decreased (Investigations) | 50 (1138)
Acidosis (Metabolism and nutrition disorders) | 8 (39)
Alkalosis (Metabolism and nutrition disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 18 (24)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 8 (13)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (6)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (5)
Hypernatremia (Metabolism and nutrition disorders) | 3 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 14 (43)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 14 (23)
Hypocalcemia (Metabolism and nutrition disorders) | 17 (48)
Hypoglycemia (Metabolism and nutrition disorders) | 8 (13)
Hypokalemia (Metabolism and nutrition disorders) | 27 (92)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3)
Hyponatremia (Metabolism and nutrition disorders) | 15 (22)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (10)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 6 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 2 (2)
Movements involuntary (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Seizure (Nervous system disorders) | 3 (3)
Delirium (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 (4)
Skin ulceration (Skin and subcutaneous tissue disorders) | 10 (10)
Hematoma (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 27 (45)
Hypotension (Vascular disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MSA states Site is unable to publish until all completed case report forms have been delivered to Sponsor, (Study Completion). Site shall have the right to publish after publication of a multi-center publication coordinated by the Sponsor or (12) mths. after Study Completion; provided, that prior to any such publication or public release of such data, Site shall furnish Sponsor with a copy of any proposed publication at least (45)days in advance of the proposed publication or presentation date.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT02553460/Prot_SAP_000.pdf